CLINICAL TRIAL: NCT07381335
Title: Comparison of the Efficacy of Phenol Neurolysis and Radiofrequency Thermocoagulation Applied to the Geniculate Nerve on Pain in Patients Undergoing Knee Arthroplasty Surgery
Brief Title: Phenol Neurolysis and Radiofrequency Thermocoagulation in Knee Arthroplasty Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Esra Ertilav, Assoc.Prof., Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025/280
Record Dates: First submitted 2026-01-20; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Radiofrequency; Arthroplasty; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): patients to whom applied radiofrequency thermocoagulation
  Interventions: Procedure: genicular nerve radiofrequency thermocoagulation and fenole neurolysis
- Group 2 (Experimental): patients to whom applied chemical neurolysis
  Interventions: Procedure: genicular nerve radiofrequency thermocoagulation and fenole neurolysis

INTERVENTIONS:
Procedure: genicular nerve radiofrequency thermocoagulation and fenole neurolysis — After visualizing the tibiofemoral joint with fluoroscopy, the potential locations of the geniculate nerves in the medial and lateral regions of the distal femur and medial tibia will be identified with fluoroscopy. A 5 cm long, 5 mm active tip RFT cannula (NeuroThermTM, Medipoint GmbH, Hamburg, Germany) is placed for each geniculate nerve using anteroposterior and lateral fluoroscopy images. Sensory stimulation at 50 Hz and motor stimulation at 2 Hz are then applied, followed by a 2 cc 0.5% bupivacaine block for each geniculate nerve. Each cannula is lesioned for 90 seconds using an 80-degree conventional RFT generator (Neurotherm NT1100 / 13001-12).
  In the phenol neurolysis group, a 22-gauge, 3.5-inch Quincke needle is advanced toward the junction of the femoral shaft and lateral condyle for the superior lateral genicular nerve. A mixture of 6 cc of 0.25% bupivacaine and 6% phenol is injected into each geniculate nerve
  Other Names: fenole neurolysis

SUMMARY:
Patients who presented to the Department of Neurology, Algology, and underwent knee arthroplasty surgery for chronic knee osteoarthritis between 2025 and 2026 and underwent radiofrequency or chemical neurolysis of the geniculate nerve due to pain will be studied in two groups. The groups will be randomly assigned by the clinician using computer-aided designation, and the patients will be allocated to the two groups. Patients in Group 1 will receive radiofrequency thermocoagulation of the geniculate nerve. Patients in Group 2 will receive phenol neurolysis of the geniculate nerve. Patients with pacemakers will be included in the phenol neurolysis group (Group 2), and patients with a phenol allergy will be included in the radiofrequency group (Group 1).

During the study, NRS and WOMAC measurements will be performed on patients in Groups 1 and 2 to assess pain intensity before the procedure and at 1, 3, and 6 months post-procedure. Neurological and musculoskeletal system examinations will be performed during routine check-ups before the procedure and at 1, 3 and 6 months after the procedure, and any developing side effects will be recorded.

DETAILED DESCRIPTION:
140 patients who underwent arthroplasty for chronic knee osteoarthritis will be evaluated in the Algology Department of the Neurology Department at Adnan Menderes University Hospitals between October 2025 and May 2026. Inclusion criteria include patients over the age of 18 who underwent arthroplasty for chronic knee osteoarthritis. Written informed consent will be obtained from all participants. Patients with severe systemic diseases, local infections, or injuries, and those allergic to any of the injection materials will be excluded. All patients will be clinically evaluated (a detailed history, including personal data, medical history, and current treatments). Procedural procedures will be performed in a sterile operating room environment. Patients are positioned supine, and a pillow is placed under the popliteal fossa to support the knee. After visualizing the tibiofemoral joint with fluoroscopy, the potential locations of the geniculate nerves in the medial and lateral regions of the distal femur and medial tibia will be identified with fluoroscopy. After sterile conditions are achieved, local anesthesia is administered both subcutaneously and transcutaneously. A 5 cm long, 5 mm active tip RFT cannula (NeuroThermTM, Medipoint GmbH, Hamburg, Germany) is placed for each geniculate nerve using anteroposterior and lateral fluoroscopy images. For the superior lateral geniculate nerve, it is advanced toward the attachment of the femoral shaft and lateral condyle, for the superior medial geniculate nerve toward the distal femoral diaphysis, and for the inferior medial geniculate nerve toward the proximal tibial diaphysis and medial tibial condyle, ensuring bone contact. The cannula is positioned midline between the diaphysis of the femur and tibia using the lateral image. Sensory stimulation at 50 Hz and motor stimulation at 2 Hz are then applied, followed by a 2 cc 0.5% bupivacaine block for each geniculate nerve. Each cannula is lesioned for 90 seconds using an 80-degree conventional RFT generator (Neurotherm NT1100 / 13001-12).

In the phenol neurolysis group, a 22-gauge, 3.5-inch Quincke needle is advanced toward the junction of the femoral shaft and lateral condyle for the superior lateral genicular nerve; toward the distal femoral diaphysis for the superior medial genicular nerve; and toward the proximal tibial diaphysis and medial tibial condyle for the inferior medial genicular nerve, ensuring bone contact. Lateral imaging confirms the cannula's position in the midline of the diaphysis of the femur and tibia. A mixture of 6 cc of 0.25% bupivacaine and 6% phenol is injected into each geniculate nerve. Post-procedure complications and side effects (infection, bleeding, neurological deficit, etc.) are recorded. Patient response will be determined according to the reduction in pain at follow-up visits at 1, 3, and 6 months after the procedure as follows: good responders will be evaluated as >50% reduction, poor responders will be evaluated as <50% reduction, or no change will be evaluated as non-responders.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria were patients over the age of 18 who had undergone arthroplasty for chronic knee osteoarthritis.Exclusion Criteria:

Exclusion Criteria:

Patients with severe systemic diseases, local infections or injuries, and those allergic to any of the injection materials were excluded from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy of both methods on knee surgery patients | 6 months
  Patients undergoing knee arthroplasty surgery for chronic knee osteoarthritis will be evaluated with the Numerical Rating Scale (NRS) before the intervention and at 1, 3, and 6 months after the procedure. A decrease in NRS of 50% or more will be considered significant.

SECONDARY OUTCOMES:
Safety of both methods on knee surgery patients | 12 months
  The aim of this study was to determine the side effects and complications of phenol and radiofrequency applications to the geniculate nerve in patients undergoing knee arthroplasty surgery for chronic knee osteoarthritis. Neurological and musculoskeletal examinations will be performed during routine checkups before and at 1, 3, and 6 months after the procedure in patients undergoing knee arthroplasty surgery for chronic knee osteoarthritis, and any developing side effects will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Esra Ertilav, Aydin, Efeler/Aydın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No